CLINICAL TRIAL: NCT02196727
Title: Evaluation of Post-operative Pain in Bascom Cleft Lift Operation Receiving Multimodal Analgesia and Spinal Saddle Block in Day Case Surgery Setting.
Brief Title: Evaluation of Postoperative Pain Following Bascom Cleft Lift Operation
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Saphana Jassim Mohamed, Consultant, Hvidovre University Hospital
Other Study IDs: BPP
Record Dates: First submitted 2014-07-18; First posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2013-05

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain; Multimodal analgesia; Bascom Cleft Lift; Day-case.
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing Bascom operation

SUMMARY:
The purpose of this study is to evaluate postoperative pain in Bascom Cleft Lift operation receiving multimodal analgesia in day-case surgery setting.

Hypothesis: Multimodal analgesia provides adequate pain relief in patients undergoing Bascom Cleft Lift operation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* ASA physical status 1 and 2
* Patient undergoing Bascom operation in prone position

Exclusion Criteria:

* Pregnancy
* Current regular use of drug belonging to the class of opioids
* Allergy/ intolerance to drugs included in multimodal analgesia regime

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing Bascom Cleft Lift operation in a day-case surgery setting
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2013-05; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) pain score (0=no pain, 10= maximum imaginable pain) | 24 hours postoperatively

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) pain score (0=no pain, 10= maximum imaginable pain) | 2 hours, 48 hours and 30 days postoperatively

OTHER OUTCOMES:
Nausea | 2 hours postoperatively
  Scale (0= non, 1= mild, 2= moderate, 3= severe)
Returning to work | 30 days
  Questionnaire: "Yes" or "No"
Returning to leisure activities | 30 days
  Questionnaire: "Yes" or "No"
Wound condition | 30 days
  Wound inspection for healing problems or infection
Vomiting | 2 hours postoperatively
  Scale (0= non, 1= mild, 2= moderate, 3= severe)

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre Univarsity Hospital, Hvidovre, Copenhagen, Denmark

REFERENCES:
- [Derived] Mohamed SJ, Kristensen BB, Lindgaard L, Bisgaard T. Acceptable effect of multimodal analgesic treatment after a Bascom cleft lift operation. Dan Med J. 2015 Jan;62(1):A4985. PMID 25557329